CLINICAL TRIAL: NCT03076840
Title: The Immediate Effect of Kinesio Tape on Hamstring Muscle Length in Female Students of University of Dammam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-PGS-2015-03-220
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Hamstring Tightness
Keywords: hamstring tightness
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio tape group (Active Comparator): treatment by: application of Kinesio tape in the hamstring muscle by using a 1 strip Y shape of (Kinesio Tex® Tape 5cm) insertion to origin technique to relieve the hamstring tightness while the muscle in stretched position for 15 second (hip flexion and knee extension and then application of the tape) with 25% stretch of the tape
  Interventions: Other: Kinesio tape
- sham tape group (Sham Comparator): treatment by: application of Kinesio tape in the hamstring muscle by using a 1 strip I shape of (Kinesio Tex® Tape 5cm) with no stretch in the hamstring musculature and the tape applied perpendicular over the upper third of the hamstring muscle while the muscle in stretched position
  Interventions: Other: Kinesio tape
- control group (No Intervention): The student in this group had no treatment in the same position of the previous groups (the hamstring muscle maintained in a stretching position for 15 second)

INTERVENTIONS:
Other: Kinesio tape — Kinesio Taping is another option for the treatment of poor hamstring extensibility, It was developed by Kenzo Kase in 1970 and gained a wide popularity by the elite athletes during the various championships and Olympic Games
  Arms: Kinesio tape group; sham tape group

SUMMARY:
The hamstring muscle is an important muscle that affect the performance of almost all activities of daily living. Since this muscle is a large muscle that pass across two major joints (the hip and knee joint), it is more susceptible to become tight and to lose its extensibility. On the other hand, there is no agreement on a standard protocol for the treatment of hamstring tightness. Kinesio tape is one of the options for treatment of hamstring muscle, it is a safe, passive and non-painful intervention, and if proven to be effective it will help individuals especially those with poor compliance and poor tolerance to painful stretching exercises. The aim of the present study is to investigate the acute effectiveness of Kinesio taping on hamstring muscles extensibility. 96 students with hamstring tightness will be recruited from the University of Dammam to participate in this prospective experimental study. All participants will be assigned randomly to either a Kinesio tape group, Sham tape group and control group. Outcome measures will be the hamstring length measurement by using active knee extension test and strength measurement for hamstring and quadriceps muscles by using a handheld dynamometer. Outcome measurement will be taken at baseline and 15 minutes after the intervention.

DETAILED DESCRIPTION:
Design:

Prospective, pre-post experimental study with three groups (Kinesio tape group, sham tape group and control group)

Setting:

This study was conducted at the laboratory of University of Dammam one session (half an hour) for each participant.

Participants:

96 students with hamstring tightness were recruited from the University of Dammam as a sample of convenience to participate in this study. These students were enrolled in the study based on the following inclusion and exclusion criteria.

Inclusion Criteria:

1. Female student with an age of 18-25 years
2. Body mass index between 18-30)
3. students with reduced hamstring length (hamstring tightness) as defined by the literature (popliteal angle less than 160 degree)

Exclusion criteria:

1. lower limb musculoskeletal pain
2. abdominal , lower limb and spinal surgery
3. pregnancy
4. previous injury or trauma to hamstring muscle, hip, knee And ankle joint
5. Skin allergy, disease or hypersensitivity
6. Low back pain or any neurological impairment in the lower extremity
7. Body mass index above 30 or below 18

Procedure:

A poster announcement was published at University of Dammam, 96 female students were recruited from a convenience sampling of students. The possible participants were approached and the idea of the research (the duration of the participation, the length of treatment session, the goal of the research, any possible risks including skin irritation or allergy from the Kinesio tape) were explained to the student. The students were instructed about dealing with any skin irritation by removing the tape and applying ice in the area for 10-15 min, students were informed that there is no compensation for any skin reaction due the Kinesio tape, although this may be less likely to happen . The students were given the chance to ask questions. If the students agree to participate in the research, they were given the consent form to read and ask a question again for any details and then they were asked to sign the consent form.

After that, the subjects were scanned for the eligibility of fitting the inclusion and exclusion criteria by the primary researcher, This was done in a safe and secured room in the laboratories of physical therapy department where the evaluation and intervention procedures were taken place. If the students fit the eligibility, then the students were undergoing a tape allergy test by applying a small piece of Kinesio tape to the patient skin for 10 minute. If the students pass this test by having no allergy reaction, then they were enrolled in the study. Students age, height, weight and body mass index(BMI) were recorded, then the students were undergo a 5 minute walking as a warming up to pre-condition the muscles before the examination. Then, hamstring length measurement, strength measurement of hamstring and quadriceps muscle were done (All students data will be coded and stored with the primary researcher through a secured password to ensure the student data confidentiality).

The outcome measures:

1. Hamstring length measurement:

   Hamstring muscle length was measured by using the active knee extension test (AKE)(Active knee extension is reliable and associated with minimal pelvic and lumber motion. Therefore, it considers a suitable and preferable test for evaluating the length of hamstring muscle. The knee extension angle (popliteal angle) was measured by using a conventional goniometer which is a reliable tool for measuring the range of motion

   The hamstring length measurement was performed with the student in a supine position with 90-degree hip flexion touching the horizontal bar apparatus.The non-tested lower limb was secured with a strap attached to the table. While the student maintains the contact between her thigh and the horizontal bar apparatus, she was asked to extend the leg as much as possible. The angle of the knee joint was measured by the researcher with a goniometer. The measurements were done three times, and the mean value were recorded
2. Hamstring and quadriceps muscle strength measurement:

The hamstring and quadriceps muscle strength were measured by the primary researcher by using the handheld dynamometer. The hamstring strength measurement was done with the student in prone position, then the student was asked to flex the knee as hard as possible while the researcher try to prevent the movement with the handheld dynamometer just proximal to the medial malleolus. The quadriceps strength measurement was done with the same procedure but from sitting position and the student was asked to extend the knee

After finishing all of the baseline outcome measures (hamstring length measurement and the strength measurement), the student were given a number and were assigned randomly to either the Kinesio tape group or the sham tape group or the control group. Each group fellow their program. The outcome measurements were repeated after 15 min at the conclusion of the treatment period

ELIGIBILITY:
Inclusion Criteria:

1. Female student with an age of 18-25 years
2. Body mass index between 18-30
3. Students with reduced hamstring length (hamstring tightness) as defined by the literature (popliteal angle less than 160 degree)

Exclusion Criteria:

1. Lower limb musculoskeletal pain
2. Abdominal, lower limb and spinal surgery
3. Pregnancy
4. Previous injury or trauma to hamstring muscle, hip, knee And ankle joint
5. Skin allergy, disease or hypersensitivity
6. Low back pain or any neurological impairment in the lower extremity
7. Body mass index above 30 or below 18

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-02-17 (Actual); Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
1- Hamstring length measurement | 5 min
  Hamstring muscle length was measured by using the active knee extension test

SECONDARY OUTCOMES:
Hamstring and quadriceps muscle strength measurement | 5 min
  The hamstring and quadriceps muscle strength were measured by the primary researcher by using the handheld dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: ennas FA Alanany, Prof, Study Director — Imam Abdulrahman Bin Faisal University
Locations (1):
- University of Dammam, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
only coded data

REFERENCES:
- [Derived] Albeshri ZS, Youssef EF. The Immediate Effect of Kinesio Tape on Hamstring Muscle Length and Strength in Female University Students: A Pre-post Experimental Study. Saudi J Med Med Sci. 2023 Jan-Mar;11(1):73-80. doi: 10.4103/sjmms.sjmms_585_22. Epub 2023 Jan 14. PMID 36909004